CLINICAL TRIAL: NCT06792344
Title: Clinical Study of CD19 Targeting Chimeric Antigen Receptor T Lymphocytes (CAR-T) in the Treatment of Refractory Systemic Sclerosis
Brief Title: Clinical Study of CD19 CAR-T in the Treatment of Refractory Systemic Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Mao Jianhua, professor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-IRB-0306-P-01
Record Dates: First submitted 2024-12-23; First posted 2025-01-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2024-12

CONDITIONS: Systemic Sclerosis (SSc)
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: CD19 CAR-T
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 CAR-T cells in the treatment of SSc (Experimental)
  Interventions: Other: anti-CD19 CAR-T cells; Drug: anti-CD19 CAR-T cells

INTERVENTIONS:
Other: anti-CD19 CAR-T cells — Intravenous injection the targeting CD19 CAR T cell
Drug: anti-CD19 CAR-T cells — CD19-targeting CAR-T cells

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety and efficacy of anti-CD19 CAR-T cells in the treatment of childhood-onset systemic sclerosis

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a type of systemic autoimmune disease characterized by skin thickening and hardening. In addition to skin involvement, it can also affect the internal organs (lungs, cardiovascular, kidney, digestive tract, etc.).

Currently there are no drugs that can affect the natural course of systemic sclerosis, and individualized treatment according to target organ involvement is usually used, glucocorticoid is used for patient combined with myositis or mixed connective tissue , and various immunosuppressants, including azathioprine, mycophenolate and cyclophosphamide, may be helpful in the treatment of interstitial lung disease. The anti-IL-6 blocker tocilizumab and the anti-fibrotic drug nitidanib have also been shown to be effective to SSC-associated interstitiallungdisease (ILD) and cardiac involvment.

Since 2019, CAR-T cell therapy has been successfully applied to autoimmune diseases. Clinical studies have demonstrated that targeted CD19 CAR-T cells hold significant therapeutic potential for SLE. These cells effectively slow down the pathological progression of SLE and can also effectively treat severe cases. Furthermore, targeted CD19 CAR-T cells are also expected to restore the immune system in SLE patients, potentially allowing them to discontinue lifelong medication and avoid serious long-term side effects of drugs like hormones and immunosuppressants. Studies have reported that CAR-T has a good therapeutic effect on a variety of autoimmune diseases such as systemic sclerosis and idiopathic inflammatory dermatomyositis.The purpose of this study is to assess the safety and efficacy of the anti-CD19 CAR-T cells in the treatment of childhood-onset refractory SSc.

ELIGIBILITY:
Inclusion Criteria:

1. Gender unlimited, age ≥5 years;
2. Meet the classification criteria for Systemic sclerosis (SSc) as defined by the 2013ACR/EULAR standards;
3. any one of the anti-nuclear antibodies or systemic sclerosis specific antibodies positive;
4. Improved Rodnan skin score (mRSS) ≥15 points (total 51 points);
5. Meet the definition of intractable disease: Glucocorticoids (≥0.5mg/kg/d) and cyclophosphamide, as well as one or more of the following immunomodulators (including antimalarial drugs, azathioprine,motecophanate, methotrexate, leflunomide, tachlimus, cyclosporine, and biologics including rituximab, Beliumab, and titacept, etc.), did not show significant remission of the disease for more than 3 months; Or meet the criteria for rapid disease progression , clinical routine treatment is ineffective, and the benefits outweigh the risks as determined by the investigator and the patient's or guardian's full and informed consent can be considered for inclusion.
6. Major organ functions were basically normal: left ventricular ejection fraction (LVEF) ≥55%, no obvious abnormality in electrocardiogram; eGFR≥30ML/min/1.73m2；AST and ALT≤3.0ULN, total bilirubin ≤2.0×ULN; SpO2≥92%, DLCO≥ 40% of predicted value, FVC≥ 50% of predicted value;
7. The subject of childbearing age has a negative urine pregnancy test result and agrees to take effective contraceptive measures during the test period until 1 year after the infusion;
8. The patient or his/her guardian agrees to participate in the clinical trial and signs an informed consent indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study

Exclusion Criteria:

（1） Severe pulmonary hypertension (PHA) (mean pulmonary pressure > 45mmHg) or other severe major organ involvement; (2) have previously received CAR T cell therapy (except those whose safety risks have been ruled out by the investigators); (3) patients with active central nervous system diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, etc.; (4) Congenital heart disease or history of acute myocardial infarction within 6 months before screening, or severe arrhythmias (including multi-source frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with a large number of pericardial effusion, serious myocarditis, etc.; Or patients with unstable vital signs who require vasoactive drugs to maintain blood pressure; (5) Active tuberculosis at the time of screening; (6) There are active infections or uncontrollable infections that require systemic treatment at the time of screening; (7) Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months before screening; Acute graft-versus-host disease (GVHD) of grade 2 or above was present within 2 weeks prior to screening; (8) Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA detection greater than the normal range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Positive for human immunodeficiency virus (HIV) antibodies; Treponema pallidum antibody positive; (9) Had received live vaccine within 4 weeks before screening; (10) Positive blood pregnancy test; (11) Patients with known malignant diseases such as tumors before screening; (12) Patients who had participated in other interventional clinical trials within 3 months before enrollment; (13) Situations in which other investigators consider it inappropriate to participate in the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | 6 months
  the Change in the modified Rodnan Skin Score (mRSS) from baseline at 6 months

SECONDARY OUTCOMES:
efficiency endpoint | the first month ,the second month ,the sixth month
  The EUSTAR activity index and combined response index (CRISS) changed after 1 month ,2 months ,6 months,12 months
PK parameter | 28 days and 90 days
  The maximum concentration (Cmax) of CD19-targeted CAR T cells in blood after infusion, the time to reach the maximum concentration (Tmax) and the area under the curve at 28 days /90 days after infusion were AUC28d/90d

CONTACTS AND LOCATIONS:
Locations (2):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, Christmas Island

IPD SHARING:
Plan to Share IPD: No